CLINICAL TRIAL: NCT00296062
Title: Dose-Dense and Dose-Intense Alternating Irinotecan/Capecitabine and Oxaliplatin/Capecitabine: Phase I in Solid Tumors and Phase II With Bevacizumab a First-Line Therapy of Advanced Colorectal Cancer
Brief Title: Dose Dense Therapy and Bevacizumab in Solid Tumors and Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial did not move to Phase II portion due to poor tolerance of treatment
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1205; U01CA062502 (NIH); P30CA043703 (NIH); CASE1205 (Other: Case Comprehensive Cancer Center); NCI-7325 (Other: CTEP/NCI)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab — Phase II: IV over 30-90 minutes on days 1 and 15 of each course.
Drug: capecitabine — Phase I: oral capecitabine twice daily on days 1-7 and 15-21.Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of capecitabine (during both odd- and even-numbered courses) until the maximum tolerated dose (MTD) is determined.Phase II:receive capecitabine (at the MTD determined in phase I(odd-numbered courses)
Drug: irinotecan hydrochloride — Phase I: irinotecan hydrochloride IV over 90 minutes on days 1 and 15 during course 1 and all subsequent odd-numbered courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.Phase II: receive capecitabine (at the MTD determined in phase I) in combination with irinotecan hydrochloride (during odd-numbered courses)
Drug: oxaliplatin — Phase I: oxaliplatin IV over 2 hours on days 1 and 15 during course 2 and all subsequent even-numbered courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Phase II: oxaliplatin (during even-numbered courses) as in phase I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, irinotecan, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also block blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of capecitabine when given together with irinotecan and oxaliplatin with or without bevacizumab and to see how well they work in treating patients with metastatic or locally advanced colorectal cancer or other solid tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
The study was originally intended to be Phase I/Phase II but it was terminated early because of toxicity of treatment and therefore never moved to the Phase II portion of the study.

OBJECTIVES:

* Determine the maximum tolerated dose (MTD) and dose-limiting toxicity of dose-dense and dose-intense capecitabine in combination with alternating full-dose irinotecan hydrochloride and oxaliplatin in patients with metastatic or locally advanced unresectable solid tumors. (phase I)
* Characterize the safety of the MTD in patients ≥ 65 years of age treated with this regimen. (phase I)
* Characterize the pharmacokinetics of this regimen in patients ≥ 65 years of age. (phase I)
* Characterize the functional status of patients ≥ 65 years of age at baseline and after study treatment, in terms of performance status, independence in activities, comorbidities, risk of malnutrition, and underlying depression. (phase I)
* Characterize the neurological status of all patients, in terms of muscle strength and sensation, at baseline and after study treatment. (phase I)
* Determine the clinical antitumor response in patients treated with this regimen. (phase I)
* Determine whether the addition of bevacizumab to dose-intense capecitabine in combination with alternating full-dose irinotecan hydrochloride and oxaliplatin as first-line treatment leads to an improved response rate in patients with metastatic colorectal cancer compared to that of published results of fluoropyrimidine/oxaliplatin, fluoropyrimidine/irinotecan/bevacizumab, and fluoropyrimidine/irinotecan regimens. (phase II)
* Determine the toxicity of bevacizumab in combination with this regimen in patients with metastatic colorectal cancer. (phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of capecitabine followed by a phase II study.

* Phase I (all solid tumor patients): Patients receive oral capecitabine twice daily on days 1-7 and 15-21. Patients also receive irinotecan hydrochloride IV over 90 minutes on days 1 and 15 during course 1 and all subsequent odd-numbered courses and oxaliplatin IV over 2 hours on days 1 and 15 during course 2 and all subsequent even-numbered courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity Cohorts of 3-6 patients receive escalating doses of capecitabine (during both odd- and even-numbered courses) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients (with at least 1 patient < 65 years of age) experience dose-limiting toxicity. At least 6 patients are treated at the MTD.
* Phase II (colorectal cancer patients): Patients receive capecitabine (at the MTD determined in phase I) in combination with irinotecan hydrochloride (during odd-numbered courses) and oxaliplatin (during even-numbered courses) as in phase I. Patients also receive bevacizumab IV over 30-90 minutes on days 1 and 15 of each course.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Phase I:

  * Histologically or cytologically confirmed solid tumor

    * Metastatic OR locally advanced unresectable disease
    * No curative therapy exists
  * Measurable or evaluable disease

    * Measurable disease is defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm with conventional techniques OR ≥ 10 mm with spiral CT scan
  * No known brain metastases
* Phase II:

  * Histologically or cytologically confirmed colorectal cancer

    * Metastatic OR locally advanced unresectable disease
  * Measurable disease (as defined in phase I)
  * No tumor involving major blood vessels
  * No evidence of CNS disease, including primary brain tumor or brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3

  * ANC < 1,500/mm^3 allowed, if in the opinion of the investigator, this represents an ethnic or racial variation of normal
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 10.0 g/dL
* Bilirubin ≤ 1.5 mg/dL
* AST/ALT ≤ 2 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio < 1.0 OR protein < 1 g by 24-hour urine collection (phase II)
* PT/INR ≤ 1.5 unless on full-dose anticoagulants (phase II)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective double-barrier contraception during and for 28 days (phase I) or 3 months (phase II) after completion of study treatment
* Fertile male patients must use effective contraception during and for 6 months after completion of study treatment
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to capecitabine, irinotecan hydrochloride, oxaliplatin, or bevacizumab
* No other uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No cardiac ischemia within the past 6 months (phase I)
* No New York Heart Association class II-IV congestive heart failure or symptomatic arrhythmia (phase II)
* No arterial thrombotic events within the past 6 months including, but not limited to, any of the following (phase II):

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina or angina requiring surgical or medical intervention
  * Myocardial infarction
* No clinically significant peripheral vascular disease (phase II)
* No history of hypertension unless well controlled (< 150/90 mm Hg) on an antihypertensive regimen (phase II)
* No evidence of bleeding diathesis or coagulopathy (phase II)
* No gastrointestinal (GI) perforation, abdominal fistula, or intra-abdominal abscess within the past 30 days (phase II)
* No significant history of bleeding events (phase II)

  * Patients with a history of significant bleeding episodes (e.g., hemoptysis or upper or lower GI bleeding) within the past 6 months are not eligible unless the source of bleeding has been resected
* No significant traumatic injury within the past 28 days (phase II)
* No serious or nonhealing wound, ulcer, or bone fracture (phase II)
* No peripheral neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered (phase I)
* At least 2 weeks since prior immunotherapy or biologic therapy and recovered (phase I)
* No prior treatment for advanced or metastatic colorectal cancer (phase II)
* More than 12 months since prior adjuvant chemotherapy and/or biologic therapy (e.g., bevacizumab or cetuximab) and recovered (phase II)
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to the only site of measurable disease unless there is measurable disease progression within the radiation port after completion of radiotherapy
* No prior radiotherapy to ≥ 20% of the bone marrow
* More than 28 days since prior major surgical procedure* or open biopsy and recovered (phase II)
* More than 14 days since prior minor surgery* and recovered (phase II)
* Concurrent full-dose anticoagulation (e.g., warfarin) allowed provided the following criteria are met (phase II):

  * Patient has an in-range INR (between 2 and 3) and is on a stable dose of oral anticoagulants or a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., known varices)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent sargramostim (GM-CSF) NOTE: *Insertion of a vascular device is not considered major or minor surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Phase II: Bevacizumab plus dose-intense capecitabine in combination with alternating full-dose irinotecan hydrochloride and oxaliplatin as first-line treatment leads to an improved response rate in patients with metastatic colorectal cancer | Courses repeat every 28 days in the absence of unacceptable toxicity.
Phase II: Determine the toxicity of bevacizumab in combination with this regimen in patients with metastatic colorectal cancer. | at end of course 2 (each course is 28 days)

SECONDARY OUTCOMES:
Phase I: Maximum tolerated dose in patients ≥ 65 years of age measured by CTC version 3.0 at end of Safety in the Elderly component of study | Receive escalating doses of capecitabine (during both odd- and even-numbered courses) until the maximum tolerated dose (MTD) is determined.

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States